CLINICAL TRIAL: NCT00667602
Title: A Phase 3, Open-Label, Randomized, Multi-Center Study to Evaluate the Safety and Immunogenicity After One or Two Doses of Novartis Meningococcal ACWY Conjugate Vaccine Administered to Healthy Infants and Toddlers
Brief Title: Safety and Immunogenicity Evaluation After One or Two Doses of Novartis Meningococcal ACWY Conjugate Vaccine in Healthy Infants and Toddlers
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Vaccines (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: V59P22; 2007-004754-82
Record Dates: First submitted 2008-04-24; First posted 2008-04-28 (Estimated); Results first posted 2013-11-07 (Estimated); Last update posted 2013-11-07 (Estimated); Status verified 2013-09

CONDITIONS: Meningococcal Meningitis
Keywords: Meningococcal; ACWY; Conjugate Vaccine; Meningitis; Toddlers; Infants; Concomitant Vaccination
MeSH Terms: conditions — Meningitis, Meningococcal; Meningitis

ARMS (3):
- MenACWY-CRM197 (2 doses) + Concomitant Vaccines (Experimental): Infants received two doses of MenACWY-CRM197 at 6 to 8 and 12 months of age and concomitant dose of PCV7 (Pneumococcal 7-valent Conjugate Vaccine) and DTPa-IPV-HepB-Hib (Diphtheria-Tetanus-acellular Pertussis, Hepatitis B, Inactivated Poliovirus and Haemophilus influenzae type b) at 12 months.
  Interventions: Biological: MenACWY-CRM197 (two doses); Biological: PCV7; Biological: DTPa-IPV-HepB-Hib
- MenACWY-CRM197 (1 dose) + Concomitant Vaccines (Experimental): Infants received one dose of MenACWY-CRM197 at 12 months of age and concomitant dose of PCV7 (Pneumococcal 7-valent Conjugate Vaccine) and DTPa-IPV-HepB-Hib (Diphtheria-Tetanus-acellular Pertussis, Hepatitis B, Inactivated Poliovirus and Haemophilus influenzae type b) at 12 months of age.
  Interventions: Biological: PCV7; Biological: DTPa-IPV-HepB-Hib; Biological: MenACWY-CRM197 (one dose)
- MenC (1 dose) + Concomitant Vaccines (Active Comparator): Infants received one dose of MenC vaccine at 12 months of age and concomitant dose of PCV7 (Pneumococcal 7-valent Conjugate Vaccine) and DTPa-IPV-HepB-Hib (Diphtheria-Tetanus-acellular Pertussis, Hepatitis B, Inactivated Poliovirus and Haemophilus influenzae type b) at 12 months of age.
  Interventions: Biological: MenC; Biological: PCV7; Biological: DTPa-IPV-HepB-Hib

INTERVENTIONS:
Biological: MenACWY-CRM197 (two doses) — Two 0.5mL doses of MenACWY conjugate vaccine (MenACWY-CRM197) was administered by intramuscular injection.
  Arms: MenACWY-CRM197 (2 doses) + Concomitant Vaccines
Biological: MenC — One 0.5mL dose of MenC vaccine was administered by intramuscular injection.
  Arms: MenC (1 dose) + Concomitant Vaccines
Biological: PCV7 — One 0.5mL dose of Pneumococcal 7-valent Conjugate Vaccine (PCV7) was administered by intramuscular injection.
Biological: DTPa-IPV-HepB-Hib — One 0.5mL dose of Combined Diphtheria-Tetanus-acellular Pertussis, Hepatitis B, Inactivated Poliovirus and Haemophilus influenzae type b (DTPa-IPV-HepB-Hib) vaccine was administered by intramuscular injection.
Biological: MenACWY-CRM197 (one dose) — One 0.5mL dose of MenACWY conjugate vaccine (MenACWY-CRM197) was administered by intramuscular injection.
  Arms: MenACWY-CRM197 (1 dose) + Concomitant Vaccines

SUMMARY:
The primary immunogenicity objective is to assess and compare the immunogenicity of one dose of MenACWY to one dose of Menjugate given to healthy toddlers at 12 months of age as measured by the percentage of subjects with serum bactericidal titers directed against N. meningitidis serogroup C ≥ 1:8 obtained in the serum bactericidal assay using human complement (hSBA).

ELIGIBILITY:
Inclusion Criteria:

* infants 6 to 8 months old inclusive, who were born after full term pregnancy and previously received three doses of both Prevenar and Infanrix-hexa vaccines at least 30 days before study entry

Exclusion Criteria:

* who previously received any meningococcal vaccine;
* who have had a previous confirmed or suspected disease caused by N. meningitidis, C. diphtheriae, C. tetani, Poliovirus, Hepatitis B, Hib, Pneumococcus or B. pertussis;
* who have had household contact with and/or intimate exposure to an individual with laboratory confirmed N. meningitidis (serogroups A, C, W135, or Y), B. pertussis, Hib, C. diphtheriae, Polio, or pneumococcal infection at any time since birth;
* Subjects with any serious, acute or chronic progressive disease

Ages: 6 Months to 8 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 662 (Actual)
Dates: Start 2008-03; Primary Completion 2009-07 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Vaccines, Study Chair — Novartis Vaccines
Locations (28):
- Germany (28):
  - Site 22, Bad Kreuznach
  - Site 38, Bad Lobenstein
  - Site 24, Balve
  - Site 3, Berlin
  - Site 27, Berlin
  - Site 20, Berlin
  - Site 26, Berlin
  - Site 13, Berlin
  - Site 31, Berlin
  - Site 25, Berlin
  - Site 15, Bönnigheim
  - Site 39, Eschwege
  - Site 32, Flensburg
  - Site 16, Frankenthal
  - Site 33, Glücksburg
  - Site 35, Hamburg
  - Site 2, Kehl
  - Site 28, Mainz
  - Site 44, Mainz
  - Site 43, München-Ramersdorf
  - Site 42, Neuhaus am Rennweg
  - Site 21, Neumünster
  - Site 9, Neumünster
  - Site 10, Oberstenfeld
  - Site 4, Stuttgart
  - Site 19, Stuttgart
  - Site 30, Weilheim I OB
  - Site 6, Wiesloch

REFERENCES:
- [Derived] Giuliani MM, Biolchi A, Keshavan P, Moriondo M, Tomei S, Santini L, Mori E, Brozzi A, Bodini M, Nieddu F, Ricci S, Mzolo T, Costantini M, Azzari C, Pellegrini M. Bactericidal antibodies against hypervirulent Neisseria meningitidis C field strains following MenC-CRM or MenACWY-CRM priming and MenACWY-CRM booster in children. Hum Vaccin Immunother. 2021 May 4;17(5):1442-1449. doi: 10.1080/21645515.2020.1833578. Epub 2020 Dec 16. PMID 33325757

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All participants enrolled were included in the trial.
Groups:
- MenACWY-CRM197 (2dose) + Concomitant Vaccines: Infants received two doses of MenACWY-CRM197 at 6-8 months and 12 months and Concomitant dose of PCV7 and DTPa-IPV-HepB-Hib at 12 months.
- MenACWY-CRM197 (1dose) + Concomitant Vaccines: Infants received one dose of MenACWY-CRM197 and Concomitant dose of PCV7 and DTPa-IPV-HepB-Hib at 12 months.
- MenC (1dose) + Concomitant Vaccines: Infants received one dose of MenC vaccine and Concomitant dose of PCV7 and DTPa-IPV-HepB-Hib at 12 months.
Period: Overall Study
Arm/Group | MenACWY-CRM197 (2dose) + Concomitant Vaccines | MenACWY-CRM197 (1dose) + Concomitant Vaccines | MenC (1dose) + Concomitant Vaccines
Started | 219 | 228 | 215
Completed | 211 | 213 | 197
Not Completed | 8 | 15 | 18
Not completed — Withdrawal by Subject | 4 | 9 | 10
Not completed — Lost to Follow-up | 4 | 5 | 6
Not completed — Administrative reason | 0 | 0 | 2
Not completed — Protocol Violation | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: As one site has been excluded, the number of subjects included in the analysis are MenACWY-CRM197 (2dose) + Concomitant Vaccines N= 196, MenACWY-CRM197 (1dose) + Concomitant Vaccines N= 205 and MenC (1dose) + Concomitant Vaccines N= 193
Groups:
- MenACWY-CRM197 (1dose) + Concomitant Vaccines: Infants received one dose of MenACWY-CRM197 at 12 months and Concomitant dose of PCV7 and DTPa-IPV-HepB-Hib at 12 months.
- MenC (1dose) + Concomitant Vaccines: Infants received one dose of MenC vaccine at 12 months and Concomitant dose of PCV7 and DTPa-IPV-HepB-Hib at 12 months.
- Total: Total of all reporting groups
Arm/Group | MenACWY-CRM197 (2dose) + Concomitant Vaccines | MenACWY-CRM197 (1dose) + Concomitant Vaccines | MenC (1dose) + Concomitant Vaccines | Total
Number analyzed (Participants) | 219 | 228 | 215 | 662
Age Continuous [Mean (Standard Deviation); unit: Days] | 208.4 (23.7) | 209.8 (22.2) | 209.3 (21.9) | 209.2 (22.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 105 | 106 | 94 | 305
  Male | 114 | 122 | 121 | 357

OUTCOME MEASURES:

1. Primary Outcome: Percentages of Subjects With Serum Bactericidal Titer ≥ 1:8 Against N.Meningitidis Serogroup C
Description: Immunogenicity of one dose of MenACWY-CRM197 vaccine to one dose of MenC vaccine one month post vaccination was measured using serum bactericidal assay with human complement (hSBA) titer ≥ 1:8 against N.meningitidis serogroup C.
Time Frame: 1 month postvaccination
Population: Analysis was done on the per-protocol (PP) set, i.e. the subjects who received the vaccine correctly; provided evaluable serum samples at the relevant time points; and had no major protocol violations as defined prior to analysis.
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | MenACWY-CRM197 (1dose) + Concomitant Vaccines | MenC (1dose) + Concomitant Vaccines
Number analyzed (Participants) | 175 | 153
Percentages of subjects | 83 [77 to 89] | 92 [86 to 95]
Statistical Analysis 1: Comparison: MenACWY-CRM197 (1dose) + Concomitant Vaccines vs MenC (1dose) + Concomitant Vaccines; The primary criterion for immunogenicity was that the lower limit of the two-sided 95% confidence interval (CI) for the difference between one dose of MenACWY-CRM197 and MenC in the percentage of subjects with hSBA ≥1:8 for serogroup C at 1 month following the 12 months vaccination was greater than -10%; Test type: Non-Inferiority or Equivalence — (PConcomitant Vaccine + MenACWY-CRM - PConcomitant Vaccine + MenC); Miettinen and Nurminen; Difference between the two groups and the associated 95% CIs were computed using the Miettinen and Nurminen method; Percentage Difference = -8, 95% CI 2-sided [-15 to -1]

2. Secondary Outcome: Percentages of Subjects With Human Serum Bactericidal Titer ≥ 1:4 Against N.Meningitidis Serogroup C
Description: Immunogenicity of one dose of MenACWY-CRM197 vaccine to one dose of MenC vaccine one month post vaccination was assessed as percentage of subjects with serum bactericidal activity using human complement (hSBA) titers ≥ 1:4 against N. meningitidis serogroup C.
Time Frame: 1 month postvaccination
Population: Analysis was done on PP set.
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | MenACWY-CRM197 (1dose) + Concomitant Vaccines | MenC (1dose) + Concomitant Vaccines
Number analyzed (Participants) | 175 | 153
Percentages of subjects | 90 [85 to 94] | 97 [93 to 99]
Statistical Analysis 1: Comparison: MenACWY-CRM197 (1dose) + Concomitant Vaccines vs MenC (1dose) + Concomitant Vaccines; The primary criterion for immunogenicity was that the lower limit of the two-sided 95% confidence interval (CI) for the difference between one dose of MenACWY-CRM197 and MenC in the percentage of subjects with hSBA ≥ 1:4 for serogroup C at 1 month following the 12 months vaccination was greater than -10%; Test type: Non-Inferiority or Equivalence — (PConcomitant Vaccine + MenACWY-CRM - PConcomitant Vaccine + MenC); Miettinen and Nurminen; Difference between the two groups and the associated 95% CIs were computed using the Miettinen and Nurminen method; Percentage difference = -7, 95% CI 2-sided [-13 to -2]

3. Secondary Outcome: Percentages of Subjects With Human Serum Bactericidal Titer ≥ 1:8 and Titer ≥ 1:4 Against N. Meningitidis Serogroups A, C, W, Y
Description: 1. Immunogenicity of two doses of MenACWY-CRM197 vaccine to one dose of MenC vaccine one month postvaccination was assessed and compared as percentages of subjects with serum bactericidal titer with human complement (hSBA) ≥ 1:8, ≥ 1:4 against N.meningitidis Serogroup C.
  2. Immunogenicity of two doses of MenACWY-CRM197 vaccine one month postvaccination was assessed as percentages of subjects with serum bactericidal titer with human complement (hSBA) ≥ 1:8, ≥ 1:4 against N.meningitidis Serogroup A, W, Y.
Time Frame: 1 month postvaccination.
Population: Analysis was done on PP set.
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | MenACWY-CRM197 (2dose) + Concomitant Vaccines | MenC (1dose) + Concomitant Vaccines
Number analyzed (Participants) | 167 | 153
Percentages of subjects
  titer ≥ 1:8, prevacc, Men A, (N=159,23) | 21 [15 to 29] | 0 [0 to 15]
  titer ≥ 1:8, postvacc, Men A (N=166,23) | 93 [88 to 97] | 0 [0 to 15]
  titer ≥ 1:8, prevacc, Men C (N=161,152) | 78 [71 to 84] | 6 [3 to 11]
  titer ≥ 1:8, postvacc, Men C (N=167,153) | 99 [96 to 100] | 92 [86 to 95]
  titer ≥ 1:8, prevacc, Men W, (N=157,23) | 68 [60 to 75] | 0 [0 to 15]
  titer ≥ 1:8, postvacc, Men W, (N=165,22) | 98 [94 to 99] | 5 [0 to 23]
  titer ≥ 1:8, prevacc, Men Y, (N=156, 23) | 69 [61 to 76] | 0 [0 to 15]
  titer ≥ 1:8, postvacc, Men Y, (N=163,22) | 96 [91 to 98] | 5 [0 to 23]
  titer ≥ 1:4, prevacc, Men A, (N=159,23) | 26 [19 to 33] | 0 [0 to 15]
  titer ≥ 1:4, postvacc, Men A, (N=166,23) | 95 [91 to 98] | 0 [0 to 15]
  titer ≥ 1:4, prevacc, Men C, (N=161,152) | 88 [81 to 92] | 7 [4 to 13]
  titer ≥ 1:4, postvacc, Men C, (N=167,153) | 99 [96 to 100] | 97 [93 to 99]
  titer ≥ 1:4, prevacc, Men W, (N=157,23) | 74 [66 to 81] | 0 [0 to 15]
  titer ≥ 1:4, postvacc, Men W, (N=165,22) | 98 [94 to 99] | 5 [0 to 23]
  titer ≥ 1:4, prevacc, Men Y, (N=156,23) | 78 [71 to 84] | 0 [0 to 15]
  titer ≥ 1:4, postvacc, Men Y, (N=163,22) | 99 [96 to 100] | 5 [0 to 23]
Statistical Analysis 1: Comparison: MenACWY-CRM197 (2dose) + Concomitant Vaccines vs MenC (1dose) + Concomitant Vaccines; Comparisons to MenC were based on the percentages of subjects with response (hSBA ≥1:8, prevaccination) to serogroup C. MenACWY was determined to be noninferior to MenC if the lower limit of the two-sided 95% CI for the difference between MenACWY and MenC in the percentage of subjects with response towards serogroup C was greater than -10%; Test type: Non-Inferiority or Equivalence — (PMenACWY - PMenC > -10%); Percentage difference; Difference between the two groups and the associated 95% CIs were computed using the Miettinen and Nurminen method; Mean Difference (Final Values) = 72, 95% CI 2-sided [64 to 79]
Statistical Analysis 2: Comparison: MenACWY-CRM197 (2dose) + Concomitant Vaccines vs MenC (1dose) + Concomitant Vaccines; Comparisons to MenC were based on the percentages of subjects with response (hSBA ≥1:8, one month postvaccination) to serogroup C. MenACWY was determined to be noninferior to MenC if the lower limit of the two-sided 95% CI for the difference between MenACWY and MenC in the percentage of subjects with response towards serogroup C was greater than -10%; Test type: Non-Inferiority or Equivalence — (PMenACWY - PMenC > -10%); Percentage difference; Difference between the two groups and the associated 95% CIs were computed using the Miettinen and Nurminen method; Mean Difference (Net) = 7, 95% CI 2-sided [3 to 13]
Statistical Analysis 3: Comparison: MenACWY-CRM197 (2dose) + Concomitant Vaccines vs MenC (1dose) + Concomitant Vaccines; Comparisons to MenC were based on the percentages of subjects with response (hSBA ≥1:4, prevaccination) to serogroup C. MenACWY was determined to be noninferior to MenC if the lower limit of the two-sided 95% CI for the difference between MenACWY and MenC in the percentage of subjects with response towards serogroup C was greater than -10%; Test type: Non-Inferiority or Equivalence — (PMenACWY - PMenC > -10%); Percentage difference; Difference between the two groups and the associated 95% CIs were computed using the Miettinen and Nurminen method; Mean Difference (Final Values) = 80, 95% CI 2-sided [73 to 86]
Statistical Analysis 4: Comparison: MenACWY-CRM197 (2dose) + Concomitant Vaccines vs MenC (1dose) + Concomitant Vaccines; Comparisons to MenC were based on the percentages of subjects with response (hSBA ≥1:4, one month postvaccination) to serogroup C. MenACWY was determined to be noninferior to MenC if the lower limit of the two-sided 95% CI for the difference between MenACWY and MenC in the percentage of subjects with response towards serogroup C was greater than -10%; Test type: Non-Inferiority or Equivalence — (PMenACWY - PMenC > -10%); Percentage difference; Difference between the two groups and the associated 95% CIs were computed using the Miettinen and Nurminen method; Mean Difference (Final Values) = 1, 95% CI 2-sided [-2 to 5]

4. Secondary Outcome: Percentages of Subjects With Human Serum Bactericidal Titer ≥ 1:8 and Titer ≥ 1:4 Against N. Meningitidis Serogroups A, W, Y
Description: Immunogenicity for one dose of MenACWY was assessed as percentages of subjects with serum bactericidal titer with human complement (hSBA) ≥ 1:8 and titer ≥ 1:4 by serogroups A, W, Y.
  Serogroup C is not shown here as it is shown in other outcome measures.
Time Frame: 1 month postvaccination.
Population: Analysis was done on PP set.
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | MenACWY-CRM197 (1dose) + Concomitant Vaccines
Number analyzed (Participants) | 175
Percentages of subjects
  titer ≥ 1:8, pre-vacc, Men A, (N=171) | 1 [0.015 to 3]
  titer ≥ 1:8, post-vacc, Men A, (N=172) | 49 [41 to 57]
  titer ≥ 1:8, pre-vacc, Men W, (N=168) | 3 [1 to 7]
  titer ≥ 1:8, post-vacc, Men W, (N=170) | 61 [53 to 68]
  titer ≥ 1:8, pre-vacc, Men Y, (N=160) | 3 [1 to 6]
  titer ≥ 1:8, post-vacc, Men Y, (N=167) | 50 [42 to 58]
  titer ≥ 1:4, pre-vacc, Men A, (N=171) | 1 [0.015 to 3]
  titer ≥ 1:4, post-vacc, Men A, (N=172) | 58 [50 to 65]
  titer ≥ 1:4, pre-vacc, Men W, (N=168) | 4 [1 to 8]
  titer ≥ 1:4, post-vacc, Men W, (N=170) | 62 [55 to 70]
  titer ≥ 1:4, pre-vacc, Men Y, (N=160) | 3 [1 to 6]
  titer ≥ 1:4, post-vacc, Men Y, (N=167) | 56 [48 to 63]

5. Secondary Outcome: Human Serum Bactericidal Activity Geometric Mean Titers After One Dose of MenACWY-CRM197 and MenC Against N.Meningitidis Serogroup C
Description: Immunogenicity of one dose of MenACWY-CRM197 vaccine to one dose of MenC vaccine one month post vaccination was assessed with geometric mean titer (GMT) of serum bactericidal assay with human complement (hSBA) against N. meningitidis serogroup C.
Time Frame: 1 month postvaccination
Population: Analysis was done on PP set.
Measure: Mean (95% Confidence Interval); unit: Titers
Arm/Group | MenACWY-CRM197 (1dose) + Concomitant Vaccines | MenC (1dose) + Concomitant Vaccines
Number analyzed (Participants) | 175 | 153
Titers
  Prevaccination (month 12) (N=174, 152) | 2.11 [1.77 to 2.51] | 2.29 [1.9 to 2.75]
  Postvaccination (month 13) (N=175,153) | 22 [18 to 28] | 31 [24 to 39]
Statistical Analysis 1: Comparison: MenACWY-CRM197 (1dose) + Concomitant Vaccines vs MenC (1dose) + Concomitant Vaccines; For comparison of the Geometric Mean Titers, prevaccination at 12 months of age, MenACWY-CRM197 was determined to be non-inferior to MenC if the lower limit of the 2-sided 95% CI for the ratio of the MenACWY-CRM197 to MenC Geometric Mean Titers for serogroup C was greater than 0.5; Test type: Non-Inferiority or Equivalence — (GMTMenACWY/GMTMenC > 0.5); ANOVA; Ratio = 0.92, 95% CI 2-sided [0.76 to 1.12]
Statistical Analysis 2: Comparison: MenACWY-CRM197 (1dose) + Concomitant Vaccines vs MenC (1dose) + Concomitant Vaccines; For comparison of the Geometric Mean Titers, one month postvaccination at 12 months of age, MenACWY-CRM197 was determined to be non-inferior to MenC if the lower limit of the 2-sided 95% CI for the ratio of the MenACWY-CRM197 to MenC Geometric Mean Titers for serogroup C was greater than 0.5; Test type: Non-Inferiority or Equivalence — (GMTMenACWY/GMTMenC > 0.5); ANOVA; Ratio = 0.73, 95% CI 2-sided [0.57 to 0.93]

6. Secondary Outcome: Human Serum Bactericidal Activity Geometric Mean Titers Against N.Meningitidis Serogroups A, W, Y
Description: Immunogenicity of one dose of MenACWY-CRM197 one month postvaccination was assessed with GMT of serum bactericidal assay with hSBA against Serogroups A, W, Y.
Time Frame: 1 month postvaccination
Population: Analysis was done on PP set.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | MenACWY-CRM197 (1dose) + Concomitant Vaccines
Number analyzed (Participants) | 172
Titers
  prevacc, Men A (N=171) | 1.99 [1.72 to 2.3]
  postvacc Men A (N=172) | 10 [7.71 to 13]
  prevacc, Men W (N=168) | 2.12 [1.71 to 2.62]
  postvacc Men W (N=170) | 14 [10 to 19]
  prevacc, Men Y (N=160) | 1.92 [1.59 to 2.32]
  postvacc Men Y (N=167) | 7.05 [5.43 to 9.15]

7. Secondary Outcome: Human Serum Bactericidal Activity Geometric Mean Titers Against N.Meningitidis Serogroups A, C, W, Y
Description: 1. The immunogenicity of two doses of MenACWY-CRM197, to a single dose of MenC was assessed and compared as measured by human Serum Bactericidal Activity Geometric Mean Titers directed against N. meningitidis serogroup C.
  2. The immunogenicity of two doses of MenACWY-CRM197, to a single dose of MenC was assessed as measured by human Serum Bactericidal Activity Geometric Mean Titers directed against N. meningitidis serogroups A, W, Y.
Time Frame: 1 month postvaccination
Population: Analysis was done on PP set.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | MenACWY-CRM197 (2dose) + Concomitant Vaccines | MenC (1dose) + Concomitant Vaccines
Number analyzed (Participants) | 167 | 153
Titers
  prevacc, Men A (N=159,23) | 3.4 [2.92 to 3.97] | 2 [1.46 to 2.73]
  postvacc Men A (N=166,23) | 75 [56 to 99] | 2.22 [1.22 to 4.04]
  prevacc, Men C (N=161,152) | 23 [19 to 28] | 2.29 [1.9 to 2.75]
  postvacc, Men C (N=167,153) | 249 [197 to 314] | 31 [24 to 39]
  prevacc, Men W (N=157,23) | 14 [11 to 17] | 1.71 [1.06 to 2.74]
  postvacc, Men W (N=165,22) | 213 [153 to 295] | 2 [0.99 to 4.03]
  prevacc, Men Y (N=156,23) | 11 [9.44 to 14] | 1.76 [1.18 to 2.63]
  postvacc, Men Y (N=163,22) | 156 [119 to 205] | 1.93 [1.06 to 3.52]
Statistical Analysis 1: Comparison: MenACWY-CRM197 (2dose) + Concomitant Vaccines vs MenC (1dose) + Concomitant Vaccines; For comparison of the GMTs (prevaccination), MenACWY was determined to be non-inferior to MenC if the lower limit of the two-sided 95% CI for the ratio of the MenACWY to MenC GMTs for serogroup C was greater than 0.5; Test type: Non-Inferiority or Equivalence — (GMTMenACWY/GMTMenjugate > 0.5); ANOVA; Ratio = 10, 95% CI 2-sided [8.43 to 13]
Statistical Analysis 2: Comparison: MenACWY-CRM197 (2dose) + Concomitant Vaccines vs MenC (1dose) + Concomitant Vaccines; For comparison of the GMTs (one month postvaccination), MenACWY was determined to be non-inferior to MenC if the lower limit of the two-sided 95% CI for the ratio of the MenACWY to MenC GMTs for serogroup C was greater than 0.5; Test type: Non-Inferiority or Equivalence — (GMTMenACWY/GMTMenjugate > 0.5); ANOVA; Ratio = 8.1, 95% CI 2-sided [6.35 to 10]

8. Secondary Outcome: Percentages of Subjects With Seroresponse Rates After One Dose of DTPa-IPV-HepB-Hib (Concomitant Vaccine)
Description: The immunogenicity of one dose of MenC to one dose of DTPa-IPV-HepB-Hib concomitant vacccine was assessed.
  For Pertussis antigens, Pertussis Toxin (PT), Filamentous Hemagglutinin (FHA) and Pertactin (PRN), the seroresponse in initially seronegative subjects (pre-vaccination antibody concentration < LLQ) is defined as post-vaccination antibody concentration >= LLQ; in initially seropositive subjects (pre-vaccination antibody concentration >=LLQ) seroresponse is defined as at least two fold increase of the pre-vaccination antibody concentration.
  Diptheria and Tetanus: primary endpoint ELISA (Enzyme-linked immunosorbent assay) >=0.1 (international unit -IU) IU/mL and the secondary endpoint is ELISA>=1.0 IU/mL.
  Polio type 1, 2 and 3: bNT (neutralization test) with >=1:8.
  HepB (HBV): primary endpoint ELISA >=10mU/mL.
  PRP-T: primary endpoint ≥ 0.15 mcg/mL and ≥ 1.00 mcg/mL.
Time Frame: 1 month postvaccination
Population: Analysis was done on PP set.
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Groups:
- MenACWY-CRM197 (1dose) + Concomitant Vaccines: Infants received one dose of MenACWY-CRM197 and concomitant dose of PCV7 and DTPa-IPV-HepBHib at 12 months.
Arm/Group | MenACWY-CRM197 (2dose) + Concomitant Vaccines | MenACWY-CRM197 (1dose) + Concomitant Vaccines | MenC (1dose) + Concomitant Vaccines
Number analyzed (Participants) | 168 | 173 | 152
Percentages of subjects
  Anti-Diphtheria Toxin ≥ 0.1 IU/mL N= (168,173,152) | 100 [98 to 100] | 100 [98 to 100] | 100 [98 to 100]
  Anti-Diphtheria Toxin ≥ 1.0 IU/mL N= (168,173,152) | 99 [96 to 100] | 98 [95 to 100] | 98 [94 to 100]
  Anti-Tetanus Toxin ≥ 0.1 IU/mL N= (168,173,152) | 100 [98 to 100] | 100 [98 to 100] | 100 [98 to 100]
  Anti-Tetanus Toxin ≥ 1.0 IU/mL N= (168,173,152) | 96 [92 to 98] | 96 [92 to 98] | 97 [93 to 99]
  FHA ELISA N=(160,169,152) | 97 [93 to 99] | 91 [86 to 95] | 96 [92 to 99]
  PRN ELISA N=(160,169,152) | 99 [97 to 100] | 98 [94 to 99] | 99 [95 to 100]
  PT ELISA N=(159,165,151) | 97 [93 to 99] | 95 [90 to 97] | 97 [92 to 99]
  polio 1 N=(157,161,148) | 100 [98 to 100] | 100 [98 to 100] | 99 [96 to 100]
  polio 2 N=157,(161,148) | 100 [98 to 100] | 99 [97 to 100] | 100 [98 to 100]
  polio 3 N=(146,151,143) | 100 [98 to 100] | 100 [98 to 100] | 100 [97 to 100]
  Hep B N=(157,161,147) | 99 [97 to 100] | 99 [96 to 100] | 99 [96 to 100]
  Anti-PRP (HIB) ≥ 0.15 μg/mL N=(168,173,151) | 100 [98 to 100] | 100 [98 to 100] | 100 [98 to 100]
  Anti-PRP (HIB) ≥ 1.0 μg/mL N=(168,173,151) | 100 [98 to 100] | 98 [95 to 100] | 99 [96 to 100]
Statistical Analysis 1: Comparison: MenACWY-CRM197 (2dose) + Concomitant Vaccines vs MenC (1dose) + Concomitant Vaccines; Immunogenicity of DTPa-IPV-HepB-Hib (Anti-Diptheria Toxin ≥0.1 IU/mL, one month postvaccination) given concomitantly with two dose of MenACWY was considered non-inferior to DTPa-IPV-HepB-Hib given concomitantly with one dose of MenC, if the lower limit of the two-sided 95% CI for the difference in the percentage of subjects with antibody response was greater than the cut-off level specified for that antigen was greater than -10%; Test type: Non-Inferiority or Equivalence — (PConcomitant Vaccine + MenACWY - PConcomitant Vaccine+MenC); Miettinen and Nurminen; Difference between the two groups and the associated 95% CIs were computed using the Miettinen and Nurminen method; Percentage difference = 0, 95% CI 2-sided [-2 to 2]
Statistical Analysis 2: Comparison: MenACWY-CRM197 (1dose) + Concomitant Vaccines vs MenC (1dose) + Concomitant Vaccines; Immunogenicity of DTPa-IPV-HepB-Hib (Anti-Diptheria Toxin ≥0.1 IU/mL, one month postvaccination) given concomitantly with one dose of MenACWY was considered non-inferior to DTPa-IPV-HepB-Hib given concomitantly with one dose of MenC, if the lower limit of the two-sided 95% CI for the difference in the percentage of subjects with antibody response was greater than the cut-off level specified for that antigen was greater than -10%; Test type: Non-Inferiority or Equivalence — (PConcomitant Vaccine + MenACWY - PConcomitant Vaccine+MenC); Miettinen and Nurminen; Difference between the two groups and the associated 95% CIs were computed using the Miettinen and Nurminen method; Percentage difference = 0, 95% CI 2-sided [-2 to 2]
Statistical Analysis 3: Comparison: MenACWY-CRM197 (2dose) + Concomitant Vaccines vs MenC (1dose) + Concomitant Vaccines; Immunogenicity of DTPa-IPV-HepB-Hib (Anti-Diptheria Toxin ≥1.0 IU/mL, one month postvaccination) given concomitantly with two dose of MenACWY was considered non-inferior to DTPa-IPV-HepB-Hib given concomitantly with one dose of MenC, if the lower limit of the two-sided 95% CI for the difference in the percentage of subjects with antibody response was greater than the cut-off level specified for that antigen was greater than -10%; Test type: Non-Inferiority or Equivalence — (PConcomitant Vaccine + MenACWY - PConcomitant Vaccine+MenC); Miettinen and Nurminen; Difference between the two groups and the associated 95% CIs were computed using the Miettinen and Nurminen method; Percentage difference = 1, 95% CI 2-sided [-3 to 5]
Statistical Analysis 4: Comparison: MenACWY-CRM197 (1dose) + Concomitant Vaccines vs MenC (1dose) + Concomitant Vaccines; Immunogenicity of DTPa-IPV-HepB-Hib (Anti-Diptheria Toxin ≥1.0 IU/mL, one month postvaccination) given concomitantly with one dose of MenACWY was considered non-inferior to DTPa-IPV-HepB-Hib given concomitantly with one dose of MenC, if the lower limit of the two-sided 95% CI for the difference in the percentage of subjects with antibody response was greater than the cut-off level specified for that antigen was greater than -10%; Test type: Non-Inferiority or Equivalence — (PConcomitant Vaccine + MenACWY - PConcomitant Vaccine+MenC); Miettinen and Nurminen; Difference between the two groups and the associated 95% CIs were computed using the Miettinen and Nurminen method; Percentage difference = 0, 95% CI 2-sided [-3 to 4]
Statistical Analysis 5: Comparison: MenACWY-CRM197 (2dose) + Concomitant Vaccines vs MenC (1dose) + Concomitant Vaccines; Immunogenicity of DTPa-IPV-HepB-Hib (Anti-Tetanus Toxin ≥ 0.1 IU/mL, one month postvaccination) given concomitantly with two dose of MenACWY was considered non-inferior to DTPa-IPV-HepB-Hib given concomitantly with one dose of MenC, if the lower limit of the two-sided 95% CI for the difference in the percentage of subjects with antibody response was greater than the cut-off level specified for that antigen was greater than -10%; Test type: Non-Inferiority or Equivalence — (PConcomitant Vaccine + MenACWY - PConcomitant Vaccine+MenC); Miettinen and Nurminen; Difference between the two groups and the associated 95% CIs were computed using the Miettinen and Nurminen method; Percentage difference = 0, 95% CI 2-sided [-2 to 2]
Statistical Analysis 6: Comparison: MenACWY-CRM197 (1dose) + Concomitant Vaccines vs MenC (1dose) + Concomitant Vaccines; Immunogenicity of DTPa-IPV-HepB-Hib (Anti-Tetanus Toxin ≥ 0.1 IU/mL, one month postvaccination) given concomitantly with one dose of MenACWY was considered non-inferior to DTPa-IPV-HepB-Hib given concomitantly with one dose of MenC, for any of the antigens, if the lower limit of the two-sided 95% CI for the difference in the percentage of subjects with antibody response was greater than the cut-off level specified for that antigen was greater than -10%; Test type: Non-Inferiority or Equivalence — (PConcomitant Vaccine + MenACWY - PConcomitant Vaccine+MenC); Miettinen and Nurminen; Difference between the two groups and the associated 95% CIs were computed using the Miettinen and Nurminen method; Percentage difference = 0, 95% CI 2-sided [-2 to 2]
Statistical Analysis 7: Comparison: MenACWY-CRM197 (2dose) + Concomitant Vaccines vs MenC (1dose) + Concomitant Vaccines; Immunogenicity of DTPa-IPV-HepB-Hib (Anti-Tetanus Toxin ≥ 1.0 IU/mL, one month postvaccination) given concomitantly with two dose of MenACWY was considered non-inferior to DTPa-IPV-HepB-Hib given concomitantly with one dose of MenC, if the lower limit of the two-sided 95% CI for the difference in the percentage of subjects with antibody response was greater than the cut-off level specified for that antigen was greater than -10%; Test type: Non-Inferiority or Equivalence — (PConcomitant Vaccine + MenACWY - PConcomitant Vaccine+MenC); Miettinen and Nurminen; Difference between the two groups and the associated 95% CIs were computed using the Miettinen and Nurminen method; Percentage difference = -2, 95% CI 2-sided [-6 to 3]
Statistical Analysis 8: Comparison: MenACWY-CRM197 (1dose) + Concomitant Vaccines vs MenC (1dose) + Concomitant Vaccines; Immunogenicity of DTPa-IPV-HepB-Hib (Anti-Tetanus Toxin ≥ 1.0 IU/mL, one month postvaccination) given concomitantly with one dose of MenACWY was considered non-inferior to DTPa-IPV-HepB-Hib given concomitantly with one dose of MenC, if the lower limit of the two-sided 95% CI for the difference in the percentage of subjects with antibody response was greater than the cut-off level specified for that antigen was greater than -10%; Test type: Non-Inferiority or Equivalence — (PConcomitant Vaccine + MenACWY - PConcomitant Vaccine+MenC); Miettinen and Nurminen; Difference between the two groups and the associated 95% CIs were computed using the Miettinen and Nurminen method; Percentage difference = -1, 95% CI 2-sided [-6 to 3]
Statistical Analysis 9: Comparison: MenACWY-CRM197 (2dose) + Concomitant Vaccines vs MenC (1dose) + Concomitant Vaccines; Immunogenicity of DTPa-IPV-HepB-Hib (polio 1, one month postvaccination), given concomitantly with two dose of MenACWY was considered non-inferior to DTPa-IPV-HepB-Hib given concomitantly with one dose of MenC, if the lower limit of the two-sided 95% CI for the difference in the percentage of subjects with antibody response was greater than the cut-off level specified for that antigen was greater than -10%; Test type: Non-Inferiority or Equivalence — (PConcomitant Vaccine + MenACWY - PConcomitant Vaccine+MenC); Miettinen and Nurminen; Difference between the two groups and the associated 95% CIs were computed using the Miettinen and Nurminen method; Percentage difference = 1, 95% CI 2-sided [-2 to 4]
Statistical Analysis 10: Comparison: MenACWY-CRM197 (1dose) + Concomitant Vaccines vs MenC (1dose) + Concomitant Vaccines; Immunogenicity of DTPa-IPV-HepB-Hib (polio 1, one month postvaccination) given concomitantly with one dose of MenACWY was considered non-inferior to DTPa-IPV-HepB-Hib given concomitantly with one dose of MenC, if the lower limit of the two-sided 95% CI for the difference in the percentage of subjects with antibody response was greater than the cut-off level specified for that antigen was greater than -10%; Test type: Non-Inferiority or Equivalence — (PConcomitant Vaccine + MenACWY - PConcomitant Vaccine+MenC); Miettinen and Nurminen; Difference between the two groups and the associated 95% CIs were computed using the Miettinen and Nurminen method; Percentage difference = 1, 95% CI 2-sided [-2 to 4]
Statistical Analysis 11: Comparison: MenACWY-CRM197 (2dose) + Concomitant Vaccines vs MenC (1dose) + Concomitant Vaccines; Immunogenicity of DTPa-IPV-HepB-Hib (polio 2, one month postvaccination) given concomitantly with two dose of MenACWY was considered non-inferior to DTPa-IPV-HepB-Hib given concomitantly with one dose of MenC, if the lower limit of the two-sided 95% CI for the difference in the percentage of subjects with antibody response was greater than the cut-off level specified for that antigen was greater than -10%; Test type: Non-Inferiority or Equivalence — (PConcomitant Vaccine + MenACWY - PConcomitant Vaccine+MenC); Miettinen and Nurminen; Difference between the two groups and the associated 95% CIs were computed using the Miettinen and Nurminen method; Percentage difference = 0, 95% CI 2-sided [-2 to 3]
Statistical Analysis 12: Comparison: MenACWY-CRM197 (1dose) + Concomitant Vaccines vs MenC (1dose) + Concomitant Vaccines; Immunogenicity of DTPa-IPV-HepB-Hib (polio 2, one month postvaccination) given concomitantly with one dose of MenACWY was considered non-inferior to DTPa-IPV-HepB-Hib given concomitantly with one dose of MenC, if the lower limit of the two-sided 95% CI for the difference in the percentage of subjects with antibody response was greater than the cut-off level specified for that antigen was greater than -10%; Test type: Non-Inferiority or Equivalence — (PConcomitant Vaccine + MenACWY - PConcomitant Vaccine+MenC); Miettinen and Nurminen; Difference between the two groups and the associated 95% CIs were computed using the Miettinen and Nurminen method; Percentage difference = -1, 95% CI 2-sided [-3 to 2]
Statistical Analysis 13: Comparison: MenACWY-CRM197 (2dose) + Concomitant Vaccines vs MenC (1dose) + Concomitant Vaccines; Immunogenicity of DTPa-IPV-HepB-Hib (polio 3, one month postvaccination) given concomitantly with two dose of MenACWY was considered non-inferior to DTPa-IPV-HepB-Hib given concomitantly with one dose of MenC, if the lower limit of the two-sided 95% CI for the difference in the percentage of subjects with antibody response was greater than the cut-off level specified for that antigen was greater than -10%; Test type: Non-Inferiority or Equivalence — (PConcomitant Vaccine + MenACWY - PConcomitant Vaccine+MenC); Miettinen and Nurminen; Difference between the two groups and the associated 95% CIs were computed using the Miettinen and Nurminen method; Percentage difference = 0, 95% CI 2-sided [-3 to 3]
Statistical Analysis 14: Comparison: MenACWY-CRM197 (1dose) + Concomitant Vaccines vs MenC (1dose) + Concomitant Vaccines; Immunogenicity of DTPa-IPV-HepB-Hib (Polio 3, one month postvaccination) given concomitantly with one dose of MenACWY was considered non-inferior to DTPa-IPV-HepB-Hib given concomitantly with one dose of MenC, if the lower limit of the two-sided 95% CI for the difference in the percentage of subjects with antibody response was greater than the cut-off level specified for that antigen was greater than -10%; Test type: Non-Inferiority or Equivalence — (PConcomitant Vaccine + MenACWY - PConcomitant Vaccine+MenC); Miettinen and Nurminen — Difference between the two groups and the associated 95% CIs were computed using the Miettinen and Nurminen method; Percentage Difference = 0, 95% CI 2-sided [-2 to 3]
Statistical Analysis 15: Comparison: MenACWY-CRM197 (2dose) + Concomitant Vaccines vs MenC (1dose) + Concomitant Vaccines; Immunogenicity of DTPa-IPV-HepB-Hib (Anti- PRP ≥ 0.15 μg/mL, one month postvaccination) given concomitantly with two dose of MenACWY was considered non-inferior to DTPa-IPV-HepB-Hib given concomitantly with one dose of MenC, if the lower limit of the two-sided 95% CI for the difference in the percentage of subjects with antibody response was greater than the cut-off level specified for that antigen was greater than -10%; Test type: Non-Inferiority or Equivalence — (PConcomitant Vaccine + MenACWY - PConcomitant Vaccine+MenC); Miettinen and Nurminen — Difference between the two groups and the associated 95% CIs were computed using the Miettinen and Nurminen method; Percentage Difference = 0, 95% CI 2-sided [-2 to 2]
Statistical Analysis 16: Comparison: MenACWY-CRM197 (1dose) + Concomitant Vaccines vs MenC (1dose) + Concomitant Vaccines; Immunogenicity of DTPa-IPV-HepB-Hib (Anti- PRP ≥ 0.15 μg/mL, one month postvaccination) given concomitantly with one dose of MenACWY was considered non-inferior to DTPa-IPV-HepB-Hib given concomitantly with one dose of MenC, if the lower limit of the two-sided 95% CI for the difference in the percentage of subjects with antibody response was greater than the cut-off level specified for that antigen was greater than -10%; Test type: Non-Inferiority or Equivalence — (PConcomitant Vaccine + MenACWY - PConcomitant Vaccine+MenC); Miettinen and Nurminen; Difference between the two groups and the associated 95% CIs were computed using the Miettinen and Nurminen method; Percentage Difference = 0, 95% CI 2-sided [-2 to 2]
Statistical Analysis 17: Comparison: MenACWY-CRM197 (2dose) + Concomitant Vaccines vs MenC (1dose) + Concomitant Vaccines; Immunogenicity of DTPa-IPV-HepB-Hib (Anti- PRP ≥ 1.0 μg/mL, one month postvaccination) given concomitantly with two dose of MenACWY was considered non-inferior to DTPa-IPV-HepB-Hib given concomitantly with one dose of MenC, if the lower limit of the two-sided 95% CI for the difference in the percentage of subjects with antibody response was greater than the cut-off level specified for that antigen was greater than -10%; Test type: Non-Inferiority or Equivalence — (PConcomitant Vaccine + MenACWY - PConcomitant Vaccine+MenC); Miettinen and Nurminen — Difference between the two groups and the associated 95% CIs were computed using the Miettinen and Nurminen method; Percentage Difference = 1, 95% CI 2-sided [-2 to 4]
Statistical Analysis 18: Comparison: MenACWY-CRM197 (1dose) + Concomitant Vaccines vs MenC (1dose) + Concomitant Vaccines; Immunogenicity of DTPa-IPV-HepB-Hib (Anti- PRP ≥ 1.0 μg/mL, one month postvaccination) given concomitantly with one dose of MenACWY was considered non-inferior to DTPa-IPV-HepB-Hib given concomitantly with one dose of MenC, if the lower limit of the two-sided 95% CI for the difference in the percentage of subjects with antibody response was greater than the cut-off level specified for that antigen was greater than -10%; Test type: Non-Inferiority or Equivalence — PConcomitant Vaccine + MenACWY - PConcomitant Vaccine+MenC); Miettinen and Nurminen; Difference between the two groups and the associated 95% CIs were computed using the Miettinen and Nurminen method; Percentage Difference = -1, 95% CI 2-sided [-4 to 2]
Statistical Analysis 19: Comparison: MenACWY-CRM197 (2dose) + Concomitant Vaccines vs MenC (1dose) + Concomitant Vaccines; Immunogenicity of DTPa-IPV-HepB-Hib (Hep B, one month postvaccination) given concomitantly with two dose of MenACWY was considered non-inferior to DTPa-IPV-HepB-Hib given concomitantly with one dose of MenC, if the lower limit of the two-sided 95% CI for the difference in the percentage of subjects with antibody response was greater than the cut-off level specified for that antigen was greater than -10%; Test type: Non-Inferiority or Equivalence — (PConcomitant Vaccine + MenACWY - PConcomitant Vaccine+MenC); Miettinen and Nurminen; Difference between the two groups and the associated 95% CIs were computed using the Miettinen and Nurminen method; Percentage Difference = 0, 95% CI 2-sided [-3 to 3]
Statistical Analysis 20: Comparison: MenACWY-CRM197 (1dose) + Concomitant Vaccines vs MenC (1dose) + Concomitant Vaccines; Immunogenicity of DTPa-IPV-HepB-Hib (Hep B, one month postvaccination) given concomitantly with one dose of MenACWY was considered non-inferior to DTPa-IPV-HepB-Hib given concomitantly with one dose of MenC, if the lower limit of the two-sided 95% CI for the difference in the percentage of subjects with antibody response was greater than the cut-off level specified for that antigen was greater than -10%; Test type: Non-Inferiority or Equivalence — (PConcomitant Vaccine + MenACWY - PConcomitant Vaccine+MenC); Miettinen and Nurminen; Difference between the two groups and the associated 95% CIs were computed using the Miettinen and Nurminen method; Percentage Difference = -1, 95% CI 2-sided [-4 to 3]

9. Secondary Outcome: Percentages of Subjects With Seroresponse Rates After One Dose of PCV7 (Concomitant Vaccine)
Description: To compare the immunogenicity of PCV7 (Pneumococcal 7-valent Conjugate)Vaccine when given concomitantly with one dose or two doses of MenACWY-CRM197 or with MenC to infants at 12 months of age.
  Seroresponse for PCV7 (PnC 4, PnC 6B, PnC 9V, PnC 14, PnC 18C, PnC 19F, PnC 23F) is defined as: a subject with primary endpoint ELISA ≥ 0.35 mcg/mL and secondary endpoint ELISA ≥ 1.0 mcg/mL.
Time Frame: 1 month postvaccination
Population: Analysis was done on PP set.
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | MenACWY-CRM197 (2dose) + Concomitant Vaccines | MenACWY-CRM197 (1dose) + Concomitant Vaccines | MenC (1dose) + Concomitant Vaccines
Number analyzed (Participants) | 163 | 168 | 150
Percentages of subjects
  PNC 4 N=(168,150) | 83 [76 to 88] | 82 [75 to 88] | 87 [81 to 92]
  PNC 6B N=(168,149) | 92 [87 to 96] | 91 [86 to 95] | 97 [93 to 99]
  PNC 9V N=(168,150) | 90 [85 to 94] | 89 [83 to 93] | 93 [88 to 97]
  PNC 14 N=(167,150) | 99 [96 to 100] | 99 [97 to 100] | 99 [96 to 100]
  PNC 18C N=(168,150) | 71 [63 to 77] | 76 [68 to 82] | 86 [79 to 91]
  PNC 19 F N=(168,150) | 81 [74 to 87] | 80 [74 to 86] | 90 [84 to 94]
  PNC 23 F N=(168,150) | 88 [82 to 92] | 89 [83 to 93] | 94 [89 to 97]
Statistical Analysis 1: Comparison: MenACWY-CRM197 (1dose) + Concomitant Vaccines vs MenC (1dose) + Concomitant Vaccines; Immunogenicity of PCV7 (PNC4, one month postvaccination)given concomitantly with one dose of MenACWY was considered non-inferior to PCV7 given concomitantly with one dose of MenC, if the lower limit of the two-sided 95% CI for the difference in the percentage of subjects with antibody response was greater than the cut-off level specified for that antigen was greater than -10%; Test type: Non-Inferiority or Equivalence — (PConcomitant Vaccine + MenACWY - PConcomitant Vaccine+MenC); Miettinen and Nurminen; Difference between the two groups and the associated 95% CIs were computed using the Miettinen and Nurminen method; Percentage difference = -5, 95% CI 2-sided [-13 to 3]
Statistical Analysis 2: Comparison: MenACWY-CRM197 (1dose) + Concomitant Vaccines vs MenC (1dose) + Concomitant Vaccines; Immunogenicity of PCV7(PNC 6B, one month postvaccination) given concomitantly with one dose of MenACWY was considered non-inferior to PCV7 given concomitantly with one dose of MenC, if the lower limit of the two-sided 95% CI for the difference in the percentage of subjects with antibody response was greater than the cut-off level specified for that antigen was greater than -10%; Test type: Non-Inferiority or Equivalence — (PConcomitant Vaccine + MenACWY - PConcomitant Vaccine+MenC); Miettinen and Nurminen; Difference between the two groups and the associated 95% CIs were computed using the Miettinen and Nurminen method; Percentage difference = -6, 95% CI 2-sided [-12 to -1]
Statistical Analysis 3: Comparison: MenACWY-CRM197 (1dose) + Concomitant Vaccines vs MenC (1dose) + Concomitant Vaccines; Immunogenicity of PCV7(PnC 9V, one month postvaccination) given concomitantly with MenACWY-CRM197 or MenC was considered non-inferior, if the lower limit of the two-sided 95% CI for the difference in the percentage of subjects with antibody response was greater than -10%; Test type: Non-Inferiority or Equivalence — (PConcomitant Vaccine + MenACWY-CRM - PConcomitant Vaccine + MenC); Miettinen and Nurminen; Difference between the two groups and the associated 95% CIs were computed using the Miettinen and Nurminen method; Percentage difference = -5, 95% CI 2-sided [-11 to 2]
Statistical Analysis 4: Comparison: MenACWY-CRM197 (1dose) + Concomitant Vaccines vs MenC (1dose) + Concomitant Vaccines; Immunogenicity of PCV7 (PNC 14, one month postvaccination) given concomitantly with one dose of MenACWY was considered non-inferior to PCV7 given concomitantly with one dose of MenC, if the lower limit of the two-sided 95% CI for the difference in the percentage of subjects with antibody response was greater than the cut-off level specified for that antigen was greater than -10%; Test type: Non-Inferiority or Equivalence — (PConcomitant Vaccine + MenACWY - PConcomitant Vaccine+MenC); Miettinen and Nurminen; Difference between the two groups and the associated 95% CIs were computed using the Miettinen and Nurminen method; Percentage difference = 0, 95% CI 2-sided [-3 to 3]
Statistical Analysis 5: Comparison: MenC (1dose) + Concomitant Vaccines; Immunogenicity of PCV7( PNC 18C, one month postvaccination) given concomitantly with one dose of MenACWY was considered non-inferior to PCV7 given concomitantly with one dose of MenC, if the lower limit of the two-sided 95% CI for the difference in the percentage of subjects with antibody response was greater than the cut-off level specified for that antigen was greater than -10%; Test type: Non-Inferiority or Equivalence — (PConcomitant Vaccine + MenACWY - PConcomitant Vaccine+MenC); Miettinen and Nurminen; Difference between the two groups and the associated 95% CIs were computed using the Miettinen and Nurminen method; Percentage difference = -10, 95% CI 2-sided [-19 to -2]
Statistical Analysis 6: Comparison: MenACWY-CRM197 (1dose) + Concomitant Vaccines vs MenC (1dose) + Concomitant Vaccines; Immunogenicity of PCV7 (PNC 19F, one month postvaccination), given concomitantly with one dose of MenACWY was considered non-inferior to PCV7 given concomitantly with one dose of MenC, if the lower limit of the two-sided 95% CI for the difference in the percentage of subjects with antibody response was greater than the cut-off level specified for that antigen was greater than -10%; Test type: Non-Inferiority or Equivalence — (PConcomitant Vaccine + MenACWY - PConcomitant Vaccine+MenC); Miettinen and Nurminen; Difference between the two groups and the associated 95% CIs were computed using the Miettinen and Nurminen method; Percentage difference = -10, 95% CI 2-sided [-17 to -2]
Statistical Analysis 7: Comparison: MenACWY-CRM197 (1dose) + Concomitant Vaccines vs MenC (1dose) + Concomitant Vaccines; Immunogenicity of PCV7 (PNC 23F, one month postvaccination) given concomitantly with one dose of MenACWY was considered non-inferior to PCV7 given concomitantly with one dose of MenC, if the lower limit of the two-sided 95% CI for the difference in the percentage of subjects with antibody response was greater than the cut-off level specified for that antigen was greater than -10%; Test type: Non-Inferiority or Equivalence — (PConcomitant Vaccine + MenACWY - PConcomitant Vaccine+MenC); Miettinen and Nurminen; Difference between the two groups and the associated 95% CIs were computed using the Miettinen and Nurminen method; Percentage difference = -5, 95% CI 2-sided [-12 to 1]
Statistical Analysis 8: Comparison: MenACWY-CRM197 (2dose) + Concomitant Vaccines vs MenC (1dose) + Concomitant Vaccines; Immunogenicity of PCV7 (PNC4, one month postvaccination) given concomitantly with two doses of MenACWY was considered non-inferior to PCV7 given concomitantly with one dose of MenC, if the lower limit of the two-sided 95% CI for the difference in the percentage of subjects with antibody response was greater than the cut-off level specified for that antigen was greater than -10%; Test type: Non-Inferiority or Equivalence — (PConcomitant Vaccine + MenACWY - PConcomitant Vaccine+MenC); Miettinen and Nurminen; Difference between the two groups and the associated 95% CIs were computed using the Miettinen and Nurminen method; Percentage difference = -5, 95% CI 2-sided [-12 to 4]
Statistical Analysis 9: Comparison: MenACWY-CRM197 (2dose) + Concomitant Vaccines vs MenC (1dose) + Concomitant Vaccines; Immunogenicity of PCV7 (PNC6B, one month postvaccination) given concomitantly with two doses of MenACWY was considered non-inferior to PCV7 given concomitantly with one dose of MenC, if the lower limit of the two-sided 95% CI for the difference in the percentage of subjects with antibody response was greater than the cut-off level specified for that antigen was greater than -10%; Test type: Non-Inferiority or Equivalence — (PConcomitant Vaccine + MenACWY - PConcomitant Vaccine+MenC); Miettinen and Nurminen; Difference between the two groups and the associated 95% CIs were computed using the Miettinen and Nurminen method; Percentage difference = -5, 95% CI 2-sided [-11 to 0]
Statistical Analysis 10: Comparison: MenACWY-CRM197 (2dose) + Concomitant Vaccines vs MenC (1dose) + Concomitant Vaccines; Immunogenicity of PCV7 (PNC 9V, one month postvaccination) given concomitantly with two doses of MenACWY was considered non-inferior to PCV7 given concomitantly with one dose of MenC, if the lower limit of the two-sided 95% CI for the difference in the percentage of subjects with antibody response was greater than the cut-off level specified for that antigen was greater than -10%; Test type: Non-Inferiority or Equivalence — (PConcomitant Vaccine + MenACWY - PConcomitant Vaccine+MenC); Miettinen and Nurminen; Difference between the two groups and the associated 95% CIs were computed using the Miettinen and Nurminen method; Percentage difference = -3, 95% CI 2-sided [-10 to 3]
Statistical Analysis 11: Comparison: MenACWY-CRM197 (2dose) + Concomitant Vaccines vs MenC (1dose) + Concomitant Vaccines; Immunogenicity of PCV7 (PNC14, one month postvaccination) given concomitantly with two doses of MenACWY was considered non-inferior to PCV7 given concomitantly with one dose of MenC, if the lower limit of the two-sided 95% CI for the difference in the percentage of subjects with antibody response was greater than the cut-off level specified for that antigen was greater than -10%; Test type: Non-Inferiority or Equivalence — (PConcomitant Vaccine + MenACWY - PConcomitant Vaccine+MenC); Miettinen and Nurminen; Difference between the two groups and the associated 95% CIs were computed using the Miettinen and Nurminen method; Percentage difference = -1, 95% CI 2-sided [-4 to 3]
Statistical Analysis 12: Comparison: MenACWY-CRM197 (2dose) + Concomitant Vaccines vs MenC (1dose) + Concomitant Vaccines; Immunogenicity of PCV7 (PNC18C, one month postvaccination) given concomitantly with two doses of MenACWY was considered non-inferior to PCV7 given concomitantly with one dose of MenC, if the lower limit of the two-sided 95% CI for the difference in the percentage of subjects with antibody response was greater than the cut-off level specified for that antigen was greater than -10%; Test type: Non-Inferiority or Equivalence — (PConcomitant Vaccine + MenACWY - PConcomitant Vaccine+MenC); Miettinen and Nurminen; Difference between the two groups and the associated 95% CIs were computed using the Miettinen and Nurminen method; Percentage difference = -15, 95% CI 2-sided [-24 to -6]
Statistical Analysis 13: Comparison: MenACWY-CRM197 (2dose) + Concomitant Vaccines vs MenC (1dose) + Concomitant Vaccines; Immunogenicity of PCV7 (PNC19F, one month postvaccination) given concomitantly with two doses of MenACWY was considered non-inferior to PCV7 given concomitantly with one dose of MenC, if the lower limit of the two-sided 95% CI for the difference in the percentage of subjects with antibody response was greater than the cut-off level specified for that antigen was greater than -10%; Test type: Non-Inferiority or Equivalence — (PConcomitant Vaccine + MenACWY - PConcomitant Vaccine+MenC); Miettinen and Nurminen; Difference between the two groups and the associated 95% CIs were computed using the Miettinen and Nurminen method; Percentage difference = -9, 95% CI 2-sided [-17 to -1]
Statistical Analysis 14: Comparison: MenACWY-CRM197 (2dose) + Concomitant Vaccines vs MenC (1dose) + Concomitant Vaccines; Immunogenicity of PCV7 (PNC23F, one month postvaccination) given concomitantly with two doses of MenACWY was considered non-inferior to PCV7 given concomitantly with one dose of MenC, if the lower limit of the two-sided 95% CI for the difference in the percentage of subjects with antibody response was greater than the cut-off level specified for that antigen was greater than -10%; Test type: Non-Inferiority or Equivalence — (PConcomitant Vaccine + MenACWY - PConcomitant Vaccine+MenC); Miettinen and Nurminen; Difference between the two groups and the associated 95% CIs were computed using the Miettinen and Nurminen method; Percentage difference = -6, 95% CI 2-sided [-13 to 0]

10. Secondary Outcome: Persistence of Immune Response Measured as Percentages of Subjects With Human Serum Bactericidal Titer ≥ 1:8 and Titer ≥ 1:4 Against N. Meningitidis Serogroup C
Description: Persistence of immune response to either one or two doses of MenACWY-CRM197 or one dose of MenC as measured by serum bactericidal assay with human complement (hSBA) titers ≥ 1:8, and titers ≥ 1:4 directed against N.meningitidis serogroup C (only for subjects enrolled in Australia).
Time Frame: 1 month postvaccination and 6-18 months postvaccination.
Population: Analysis was done on PP set (persistence subgroup).
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | MenACWY-CRM197 (2dose) + Concomitant Vaccines | MenACWY-CRM197 (1dose) + Concomitant Vaccines | MenC (1dose) + Concomitant Vaccines
Number analyzed (Participants) | 17 | 14 | 13
Percentages of subjects
  hSBA ≥ 1:8, postvacc, Men C. N=(17,14,13) | 100 [80 to 100] | 86 [57 to 98] | 92 [64 to 100]
  hSBA ≥ 1:8, perisistence, Men C. N=(17,14,13) | 71 [44 to 90] | 64 [35 to 87] | 54 [25 to 81]
  hSBA ≥ 1:4, postvacc, Men C. N=(17,14,13) | 100 [80 to 100] | 93 [66 to 100] | 100 [75 to 100]
  hSBA ≥ 1:4, persistence, Men C. N=(17,14,13) | 76 [50 to 93] | 71 [42 to 92] | 77 [46 to 95]

11. Secondary Outcome: Persistence of Immune Response Measured as Percentages of Subjects With Human Serum Bactericidal Titer ≥ 1:8 ,and Titer ≥ 1:4 Against N. Meningitidis Serogroups A, W, Y
Description: Persistence of immune response to either one or two doses of MenACWY-CRM197 or one dose of MenC as measured by serum bactericidal assay with human complement (hSBA) titer ≥ 1:8 and titer ≥ 1:4 directed against N. meningitidis serogroups A, W and Y (only for subjects enrolled in Australia).
Time Frame: 1 month postvaccination 6-18 months postvaccination
Population: Analysis was done on PP set (persistence subset).
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | MenACWY-CRM197 (2dose) + Concomitant Vaccines | MenACWY-CRM197 (1dose) + Concomitant Vaccines
Number analyzed (Participants) | 17 | 14
Percentages of subjects
  hSBA ≥ 1:8, postvacc, Men A (N=17,14) | 88 [64 to 99] | 42 [15 to 72]
  hSBA ≥ 1:8, persistence, Men A (N=16,14) | 31 [11 to 59] | 7 [0 to 34]
  hSBA ≥ 1:4, post-vacc, Men A (N=17,12) | 100 [80 to 100] | 50 [21 to 79]
  hSBA ≥ 1:4, persistence, Men A (N=16,14) | 38 [15 to 65] | 14 [2 to 43]
  hSBA ≥ 1:8, postvacc, Men W (N=17,12) | 100 [80 to 100] | 67 [35 to 90]
  hSBA ≥ 1:8, persistence, Men W (N=16,14) | 75 [48 to 93] | 71 [42 to 92]
  hSBA ≥ 1:4, postvacc, Men W (N=17,13) | 86 [57 to 98] | 0 [0 to 25]
  hSBA ≥ 1:4, persistence, Men W (N=16,14) | 88 [62 to 98] | 71 [42 to 92]
  hSBA ≥ 1:8, postvacc, Men Y (N=17,12) | 100 [80 to 100] | 33 [10 to 65]
  hSBA ≥ 1:8, persistence, Men Y (N=14,14) | 79 [49 to 95] | 79 [49 to 95]
  hSBA ≥ 1:4, postvacc, Men Y (N=17,12) | 100 [80 to 100] | 50 [21 to 79]
  hSBA ≥ 1:4, persistence, Men Y (N=14,14) | 86 [57 to 98] | 93 [66 to 100]

12. Secondary Outcome: Persistence of Human Serum Bactericidal Activity Geometric Mean Titers Against N.Meningitidis Serogroup C
Description: Persistence of immunogenicity of either one or two doses of MenACWY or one dose of MenC as measured by human serum bactericidal activity geometric mean titers directed against N.meningitidis serogroup C (only for subjects enrolled in Australia).
Time Frame: 1 month postvaccination and 6-18 months postvaccination.
Population: Analysis was done on PP set (subjects enrolled in Australia).
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Groups:
- MenC(1dose) + Concomitant Vaccines: Infants received one dose of MenC vaccine and Concomitant dose of PCV7 and DTPa-IPV-HepB-Hib at 12 months.
Arm/Group | MenACWY-CRM197 (2dose) + Concomitant Vaccines | MenACWY-CRM197 (1dose) + Concomitant Vaccines | MenC(1dose) + Concomitant Vaccines
Number analyzed (Participants) | 17 | 14 | 13
Titers
  Month 13 | 241 [139 to 419] | 36 [19 to 66] | 30 [16 to 56]
  6 - 18 months after month 12 | 15 [7.45 to 29] | 12 [5.65 to 25] | 8.95 [4.15 to 19]

13. Secondary Outcome: Persistence of Human Serum Bactericidal Activity Geometric Mean Titers Against N.Meningitidis Serogroups A, W, Y
Description: Immunogenicity of two doses of MenACWY to one dose of MenACWY as measured by hSBA GMTs directed against N.meningitidis serogroups A, W, Y (only for subjects enrolled in Australia).
Time Frame: 6-18 months postvaccination.
Population: Analysis was done on PP set (only for subjects enrolled in Australia).
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | MenACWY-CRM197 (2dose) + Concomitant Vaccines | MenACWY-CRM197 (1dose) + Concomitant Vaccines
Number analyzed (Participants) | 17 | 14
Titers
  Month 12, Ser A (N= 17, 12) | 47 [26 to 86] | 6.69 [3.28 to 14]
  6 - 18 months after Month 12, Ser A (N=16,14) | 4.41 [2.78 to 7] | 2.78 [1.7 to 4.56]
  Month 12, Ser W (N= 17, 12) | 180 [95 to 340] | 13 [6.26 to 28]
  6 - 18 months after Month 12, Ser W (N=16,14) | 20 [10 to 39] | 20 [9.77 to 42]
  Month 12, Ser Y (N= 17, 12) | 151 [93 to 246] | 5.13 [2.87 to 9.17]
  6 - 18 months after Month 12, Ser Y (N=14,14) | 22 [12 to 38] | 16 [9.15 to 28]

14. Secondary Outcome: Percentages of Subjects With Rabbit Serum Bactericidal ≥ 1:8, ≥ 1:128 and Four Fold Rise Against N.Meningitidis Serogroup C
Description: 1. Immunogenicity of one dose of MenACWY-CRM197 vaccine to one dose of MenC vaccine one month post vaccination was assessed as percentages of subjects with serum bactericidal titer with rabbit complement (rSBA) ≥ 1:8, ≥ 1:128, and four fold rise in titer against N.meningitidis Serogroup C.
  2. Immunogenicity of two doses of MenACWY-CRM197 vaccine to one dose of MenC vaccine one month post vaccination was assessed as percentages of subjects with serum bactericidal titer with rabbit complement (rSBA) ≥ 1:8, ≥ 1:128, and four fold rise in titer against N.meningitidis Serogroup C.
Time Frame: 1 month postvaccination.
Population: Analysis was done on PP set.
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | MenACWY-CRM197 (2dose) + Concomitant Vaccines | MenACWY-CRM197 (1dose) + Concomitant Vaccines | MenC (1dose) + Concomitant Vaccines
Number analyzed (Participants) | 156 | 157 | 145
Percentages of subjects
  rSBA titer ≥ 1:8, prevacc (N=140,140,139) | 72 [64 to 79] | 4 [1 to 8] | 1 [0 to 5]
  rSBA titer ≥ 1:8, postvacc (N=156,157,145) | 98 [94 to 100] | 92 [86 to 96] | 97 [92 to 99]
  rSBA titer ≥ 1:128, prevacc (N=140,140,139) | 31 [23 to 39] | 1 [0.018 to 4] | 0 [0 to 3]
  rSBA titer ≥ 1:128, postvacc (N=156,157,145) | 92 [87 to 96] | 75 [68 to 82] | 88 [82 to 93]
  four fold rise (N=132,140,139) | 86 [79 to 92] | 91 [86 to 95] | 96 [92 to 99]
Statistical Analysis 1: Comparison: MenACWY-CRM197 (2dose) + Concomitant Vaccines vs MenC (1dose) + Concomitant Vaccines; For the comparisons to MenC based on percentages of subjects with response (rSBA ≥1:8, prevaccination), MenACWY-CRM197 was determined to be non-inferior to MenC if the lower limit of the two-sided 95% CI for the difference between MenACWY-CRM197 and MenC in the percentage of subjects with response against serogroup C was greater than -10%; Test type: Non-Inferiority or Equivalence — (PConcomitant Vaccine + MenACWY-CRM - PConcomitant Vaccine + MenC); Miettinen and Nurminen; Difference between the two groups and the associated 95% CIs were computed using the Miettinen and Nurminen method; Percentage difference = 71, 95% CI 2-sided [63 to 78]
Statistical Analysis 2: Comparison: MenACWY-CRM197 (2dose) + Concomitant Vaccines vs MenC (1dose) + Concomitant Vaccines; For the comparisons to MenC based on percentages of subjects with response (rSBA ≥1:8, one month postvaccination), MenACWY-CRM197 was determined to be non-inferior to MenC if the lower limit of the two-sided 95% CI for the difference between MenACWY-CRM197 and MenC in the percentage of subjects with response against serogroup C was greater than -10%; Test type: Non-Inferiority or Equivalence — (PConcomitant Vaccine + MenACWY-CRM - PConcomitant Vaccine + MenC); Miettinen and Nurminen; Difference between the two groups and the associated 95% CIs were computed using the Miettinen and Nurminen method; Percentage difference = 2, 95% CI 2-sided [-3 to 6]
Statistical Analysis 3: Comparison: MenACWY-CRM197 (1dose) + Concomitant Vaccines vs MenC (1dose) + Concomitant Vaccines; [analysis description as in outcome 14, analysis 1]; Test type: Non-Inferiority or Equivalence — (PConcomitant Vaccine + MenACWY-CRM - PConcomitant Vaccine + MenC); Miettinen and Nurminen; Difference between the two groups and the associated 95% CIs were computed using the Miettinen and Nurminen method; Percentage difference = 2, 95% CI 2-sided [-2 to 7]
Statistical Analysis 4: Comparison: MenACWY-CRM197 (1dose) + Concomitant Vaccines vs MenC (1dose) + Concomitant Vaccines; [analysis description as in outcome 14, analysis 2]; Test type: Non-Inferiority or Equivalence — (PConcomitant Vaccine + MenACWY-CRM - PConcomitant Vaccine + MenC); Miettinen and Nurminen; Difference between the two groups and the associated 95% CIs were computed using the Miettinen and Nurminen method; Percentage difference = -5, 95% CI 2-sided [-11 to 1]
Statistical Analysis 5: Comparison: MenACWY-CRM197 (2dose) + Concomitant Vaccines vs MenC (1dose) + Concomitant Vaccines; For the comparisons to MenC based on percentages of subjects with response (rSBA ≥1:128, prevaccination), MenACWY-CRM197 was determined to be non-inferior to MenC if the lower limit of the two-sided 95% CI for the difference between MenACWY-CRM197 and MenC in the percentage of subjects with response against serogroup C was greater than -10%; Test type: Non-Inferiority or Equivalence — (PConcomitant Vaccine + MenACWY-CRM - PConcomitant Vaccine + MenC); Miettinen and Nurminen; Difference between the two groups and the associated 95% CIs were computed using the Miettinen and Nurminen method; Percentage difference = 31, 95% CI 2-sided [24 to 39]
Statistical Analysis 6: Comparison: MenACWY-CRM197 (2dose) + Concomitant Vaccines vs MenC (1dose) + Concomitant Vaccines; For the comparisons to MenC based on percentages of subjects with response (rSBA ≥1:128, one month postvaccination), MenACWY-CRM197 was determined to be non-inferior to MenC if the lower limit of the two-sided 95% CI for the difference between MenACWY-CRM197 and MenC in the percentage of subjects with response against serogroup C was greater than -10%; Test type: Non-Inferiority or Equivalence — (PConcomitant Vaccine + MenACWY-CRM - PConcomitant Vaccine + MenC); Miettinen and Nurminen; Difference between the two groups and the associated 95% CIs were computed using the Miettinen and Nurminen method; Percentage difference = 1, 95% CI 2-sided [-2 to 4]
Statistical Analysis 7: Comparison: MenACWY-CRM197 (1dose) + Concomitant Vaccines vs MenC (1dose) + Concomitant Vaccines; [analysis description as in outcome 14, analysis 5]; Test type: Non-Inferiority or Equivalence — PConcomitant Vaccine + MenACWY-CRM - PConcomitant Vaccine + MenC); Miettinen and Nurminen; Difference between the two groups and the associated 95% CIs were computed using the Miettinen and Nurminen method; Percentage Difference = 4, 95% CI 2-sided [-3 to 11]
Statistical Analysis 8: Comparison: MenACWY-CRM197 (1dose) + Concomitant Vaccines vs MenC (1dose) + Concomitant Vaccines; [analysis description as in outcome 14, analysis 6]; Test type: Non-Inferiority or Equivalence — PConcomitant Vaccine + MenACWY-CRM - PConcomitant Vaccine + MenC); Miettinen and Nurminen; Difference between the two groups and the associated 95% CIs were computed using the Miettinen and Nurminen method; Percentage Difference = -13, 95% CI 2-sided [-22 to -5]
Statistical Analysis 9: Comparison: MenACWY-CRM197 (2dose) + Concomitant Vaccines vs MenC (1dose) + Concomitant Vaccines; For the comparisons to MenC based on percentages of subjects with response (four-fold rise in titers), MenACWY-CRM197 was determined to be non-inferior to MenC if the lower limit of the two-sided 95% CI for the difference between MenACWY-CRM197 and MenC in the percentage of subjects with response against serogroup C was greater than -10%; Test type: Non-Inferiority or Equivalence — PConcomitant Vaccine + MenACWY-CRM - PConcomitant Vaccine + MenC); Miettinen and Nurminen; Difference between the two groups and the associated 95% CIs were computed using the Miettinen and Nurminen method; Percentage Difference = -10, 95% CI 2-sided [-17 to -4]
Statistical Analysis 10: Comparison: MenACWY-CRM197 (1dose) + Concomitant Vaccines vs MenC (1dose) + Concomitant Vaccines; [analysis description as in outcome 14, analysis 9]; Test type: Non-Inferiority or Equivalence — PConcomitant Vaccine + MenACWY-CRM - PConcomitant Vaccine + MenC); Miettinen and Nurminen; Difference between the two groups and the associated 95% CIs were computed using the Miettinen and Nurminen method; Percentage Difference = -5, 95% CI 2-sided [-11 to 1]

15. Secondary Outcome: Percentages of Subjects With Rabbit Serum Bactericidal ≥ 1:8, ≥ 1:128, and Four Fold Rise Against N.Meningitidis Serogroup A, W, Y
Description: 1. Immunogenicity of one dose of MenACWY-CRM197 vaccine to one dose of MenC vaccine one month post vaccination was assessed as percentages of subjects with serum bactericidal titer with rabbit complement (rSBA) ≥ 1:8, ≥ 1:128, and four fold rise in titer against N.meningitidis Serogroup A, W, Y.
  2. Immunogenicity of two doses of MenACWY-CRM197 vaccine to one dose of MenC vaccine one month post vaccination was assessed as percentages of subjects with serum bactericidal titer with rabbit complement (rSBA) ≥ 1:8, ≥ 1:128, and four fold rise in titer against N.meningitidis Serogroup A, W, Y.
Time Frame: 1 month postvaccination.
Population: Analysis was done on PP set.
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | MenACWY-CRM197 (2dose) + Concomitant Vaccines | MenACWY-CRM197 (1dose) + Concomitant Vaccines
Number analyzed (Participants) | 76 | 83
Percentages of subjects
  rSBA titer ≥ 1:128, Men A | 100 [95 to 100] | 98 [92 to 100]
  rSBA titer ≥ 1:128, Men W | 96 [89 to 99] | 93 [85 to 97]
  rSBA titer ≥ 1:128, Men Y | 89 [80 to 95] | 86 [76 to 92]
  rSBA titer ≥ 1:8, Men A | 100 [95 to 100] | 98 [92 to 100]
  rSBA titer ≥ 1:8, Men W | 100 [95 to 100] | 95 [88 to 99]
  rSBA titer ≥ 1:8, Men Y | 97 [91 to 100] | 88 [79 to 94]
  Four Fold Rise of rSBA titer, Men A | 75 [64 to 85] | 95 [88 to 99]
  Four Fold Rise of rSBA titer, Men W | 95 [86 to 99] | 95 [87 to 99]
  Four Fold Rise of rSBA titer, Men Y | 91 [75 to 98] | 87 [74 to 95]

16. Secondary Outcome: Rabbit Serum Bactericidal Activity Geometric Mean Titers Against N.Meningitidis Serogroup C
Description: 1. Immunogenicity of one dose of MenACWY-CRM197 to one dose of MenC vaccine at 12 months of age was assessed with geometric mean titer (GMT) of serum bactericidal assay with rabbit complement (rSBA) against Serogroup C.
  2. Immunogenicity of two doses of MenACWY-CRM197 to one dose of MenC vaccine at 6 to 8 and 12 months of age was assessed with geometric mean titer (GMT) of serum bactericidal assay with rabbit complement (rSBA) against Serogroup C.
Time Frame: 1 month postvaccination.
Population: Analysis was done on PP set.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | MenACWY-CRM197 (2dose) + Concomitant Vaccines | MenACWY-CRM197 (1dose) + Concomitant Vaccines | MenC (1dose) + Concomitant Vaccines
Number analyzed (Participants) | 156 | 157 | 145
Titers
  GMT, prevacc (N=140,140,139) | 26 [21 to 33] | 2.22 [1.76 to 2.8] | 2.03 [1.62 to 2.54]
  GMT, postvacc (N=156,157,145) | 353 [260 to 479] | 131 [98 to 176] | 266 [197 to 359]
Statistical Analysis 1: Comparison: MenACWY-CRM197 (2dose) + Concomitant Vaccines vs MenC (1dose) + Concomitant Vaccines; For comparison of the Geometric Mean Titers at one month postvaccination at 12 months of age, MenACWY-CRM197 was determined to be non-inferior to MenC if the lower limit of the 2-sided 95% CI for the ratio of the MenACWY-CRM197 to MenC Geometric Mean Titers for serogroup C was greater than 0.5; Test type: Non-Inferiority or Equivalence — (PConcomitant Vaccine + MenACWY-CRM - PConcomitant Vaccine + MenC); ANOVA; Ratio = 1.33, 95% CI 2-sided [0.96 to 1.83]

17. Secondary Outcome: Rabbit Serum Bactericidal Activity Geometric Mean Titers Against N.Meningitidis Serogroup A, W, Y
Description: 1. Immunogenicity of one dose of MenACWY-CRM197 to one dose of MenC vaccine at 12 months of age was assessed with GMT of SBA with rabbit complement (rSBA) against Serogroup A, W, Y.
  2. Immunogenicity of two doses of MenACWY-CRM197 to one dose of MenC vaccine at 6 to 8 and 12 months of age was assessed with geometric mean titer (GMT) of serum bactericidal assay with rabbit complement (rSBA) against Serogroup A, W, Y.
Time Frame: 1 month postvaccination.
Population: Analysis was done on PP set.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | MenACWY-CRM197 (2dose) + Concomitant Vaccines | MenACWY-CRM197 (1dose) + Concomitant Vaccines
Number analyzed (Participants) | 76 | 83
Titers
  GMT, prevacc, Men A (N=73,82) | 281 [134 to 587] | 6.83 [3.34 to 14]
  GMT, postvacc, Men A | 3136 [2013 to 4886] | 3258 [2113 to 5022]
  GMT, prevacc, Men W (N=59,75) | 20 [12 to 33] | 2.32 [1.46 to 3.69]
  GMT, postvacc, Men W | 708 [421 to 1191] | 1306 [786 to 2169]
  GMT, prevacc, Men Y (N=32,49) | 22 [12 to 40] | 2.4 [1.42 to 4.06]
  GMT, postvacc, Men Y (N=76,81) | 574 [320 to 1028] | 598 [336 to 1066]

18. Secondary Outcome: Number of Subjects Who Reported Solicited Local and Systemic Reactions (Day 1 to Day 7 Postvaccination), After Any Vaccination
Description: Safety was assessed as the number of subjects who reported solicited local reactions from day 1 to day 7 postvaccination for all the three vaccination groups.
  safety was assessed as the number of subjects who reported solicited systemic reactions from day 1 to day 7 Following the Month 12 vaccination in all three vaccination groups
Time Frame: From day 1 to day 7 postvaccination
Population: Analysis was done on the safety dataset, i.e. the subjects in the exposed population who provided postvaccination safety data.
Measure: Number; unit: Number of subjects
Arm/Group | MenACWY-CRM197 (2dose) + Concomitant Vaccines | MenACWY-CRM197 (1dose) + Concomitant Vaccines | MenC (1dose) + Concomitant Vaccines
Number analyzed (Participants) | 195 | 192 | 179
Number of subjects
  Any Local N=(195,192,179) | 130 | 131 | 135
  Tenderness (MenACWY-CRM197/MenC)N=(194,192,178) | 57 | 65 | 44
  Erythema (MenACWY-CRM197/MenC) N=(194,192,178) | 94 | 62 | 64
  Induration (MenACWY-CRM197/MenC) N=(194,192,178) | 53 | 24 | 43
  Tenderness (DTPa-IPV-HepB-Hib) N=(189,190,176) | 62 | 83 | 73
  Erythema (DTPa-IPV-HepB-Hib)B N=(189,190,176) | 80 | 81 | 96
  Induration (DTPa-IPV-HepB-Hib) N=(189,190,176) | 62 | 66 | 81
  Tenderness (PCV7) N=(189,190,176) | 58 | 68 | 60
  Erythema (PCV7) N=(189,190,176) | 71 | 68 | 77
  Induration (PCV7) N=(189,190,176) | 50 | 50 | 59
  Any Systemic reactions N=(195,192,179) | 173 | 149 | 150
  Change in eating habits N=(189, 191,177) | 62 | 66 | 49
  Sleepiness N=(191,191,179) | 93 | 99 | 94
  Persistent crying N=(189,191,177) | 77 | 93 | 76
  Irritability N=(191,191,179) | 67 | 68 | 73
  Vomiting N=(191,191,179) | 10 | 18 | 16
  Diarrhoea N=(191,191,179) | 26 | 41 | 42
  Rash N=(191,191,179) | 7 | 17 | 7
  Fever ≥ 38.5C N=(191,192,179) | 54 | 62 | 50
  Others N=(195,192,179) | 64 | 62 | 62
  Analgesic-Antipyretic medication N=(191,192,179) | 58 | 62 | 62

ADVERSE EVENTS:
Time Frame: Solicited Adverse Events (AEs) were collected from Days 1-7 after any vaccination. Other AEs and Serious AEs were collected from days 1 to 180.
Description: Data collected from one site were not included in the data analysis for outcome measures and the AE section.
Arm/Group | MenACWY-CRM197 (2dose) + Concomitant Vaccines | MenACWY-CRM197 (1dose) + Concomitant Vaccines | MenC (1dose) + Concomitant Vaccines
Serious Adverse Events (participants affected / at risk) | 13/195 | 19/192 | 12/179
Other Adverse Events (participants affected / at risk) | 192/195 | 184/192 | 170/179
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MenACWY-CRM197 (2dose) + Concomitant Vaccines (N=195) | MenACWY-CRM197 (1dose) + Concomitant Vaccines (N=192) | MenC (1dose) + Concomitant Vaccines (N=179)
Lymphadenitis (Blood and lymphatic system disorders) | 0 | 1 | 0
Amphthous stomatitis (Gastrointestinal disorders) | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0
Intussusception (Gastrointestinal disorders) | 1 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 2 | 0
Hyperpyrexia (General disorders) | 1 | 1 | 0
Food Allergy (Immune system disorders) | 0 | 0 | 1
Appendicitis (Infections and infestations) | 0 | 1 | 0
Bronchitis (Infections and infestations) | 2 | 3 | 0
Croup infectious (Infections and infestations) | 0 | 0 | 1
Febrile infection (Infections and infestations) | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 3 | 4 | 4
Influenza (Infections and infestations) | 1 | 1 | 0
Malaria (Infections and infestations) | 1 | 0 | 0
Otitis media (Infections and infestations) | 0 | 1 | 3
Pneumonia (Infections and infestations) | 0 | 1 | 0
Pneumonia respiratory syncytial viral (Infections and infestations) | 1 | 1 | 0
Sepsis (Infections and infestations) | 0 | 0 | 1
Tonsillitis (Infections and infestations) | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 1 | 0
Viral infection (Infections and infestations) | 0 | 0 | 1
Accidental exposure (Injury, poisoning and procedural complications) | 0 | 1 | 0
Concussion (Injury, poisoning and procedural complications) | 1 | 2 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 1 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 2 | 0 | 1
Neuroblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Febrile convulsion (Nervous system disorders) | 0 | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | MenACWY-CRM197 (2dose) + Concomitant Vaccines (N=195) | MenACWY-CRM197 (1dose) + Concomitant Vaccines (N=192) | MenC (1dose) + Concomitant Vaccines (N=179)
Conjunctivitis (Eye disorders) | 36 | 15 | 18
Diarrhoea (Gastrointestinal disorders) | 54 | 44 | 44
Enteritis (Gastrointestinal disorders) | 13 | 4 | 5
Teething (Gastrointestinal disorders) | 21 | 6 | 7
Vomiting (Gastrointestinal disorders) | 38 | 24 | 19
Injection site erythema (General disorders) | 110 | 102 | 110
Injection site induration (General disorders) | 86 | 82 | 104
Injection site pain (General disorders) | 90 | 97 | 84
Irritability (General disorders) | 85 | 68 | 73
Pyrexia (General disorders) | 127 | 111 | 102
Bronchitis (Infections and infestations) | 47 | 29 | 29
Gastroenteritis (Infections and infestations) | 22 | 14 | 12
Nasopharyngitis (Infections and infestations) | 19 | 14 | 14
Otitis media (Infections and infestations) | 33 | 22 | 21
Rhinitis (Infections and infestations) | 24 | 7 | 8
Upper respiratory tract infection (Infections and infestations) | 67 | 31 | 29
Viral infection (Infections and infestations) | 38 | 26 | 26
Crying (Nervous system disorders) | 100 | 93 | 76
Somnolence (Nervous system disorders) | 126 | 99 | 94
Eating disorder (Psychiatric disorders) | 87 | 66 | 49
Cough (Respiratory, thoracic and mediastinal disorders) | 25 | 11 | 10
Dermatitis Diaper (Skin and subcutaneous tissue disorders) | 24 | 20 | 9
Rash (Skin and subcutaneous tissue disorders) | 28 | 24 | 7

LIMITATIONS AND CAVEATS:
GCP compliance issues were identified at one site, data collected for this site were not used in this data posting.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days